CLINICAL TRIAL: NCT03103412
Title: Study 0146: A Phase 1a, Double-Blinded, Randomized, Placebo Controlled, Single Ascending Dose (SAD) Study to Evaluate the Safety, Tolerability, and Systemic Exposure of TD-3504 in Healthy Subjects and Subjects With Ulcerative Colitis (UC)
Brief Title: TD-3504 SAD in Healthy Subjects and Subjects With Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0146
Record Dates: First submitted 2017-03-24; First posted 2017-04-06 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Active Mild Ulcerative Colitis, Active Moderate Ulcerative Colitis, Healthy Subjects
Keywords: Active Mild Ulcerative Colitis, Active Moderate Ulcerative Colitis, Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TD-3504 Low-Dose (Experimental): 6 healthy subjects and 6 ulcerative colitis subjects will be randomized to receive low-dose TD-3504 and low-dose of 15N2-tofacitinib orally single dose.
  Interventions: Drug: TD-3504; Drug: 15N2-tofacitinib
- TD-3504 Mid-Dose (Experimental): 6 healthy subjects will be randomized to receive mid-dose TD-3504 and low-dose of 15N2-tofacitinib orally single dose.
  Interventions: Drug: TD-3504; Drug: 15N2-tofacitinib
- TD-3504 High-Dose (Experimental): 6 healthy subjects will be randomized to receive high-dose TD-3504 and low-dose of 15N2-tofacitinib orally single dose.
  Interventions: Drug: TD-3504; Drug: 15N2-tofacitinib
- Placebo (Placebo Comparator): 6 healthy subjects and 2 ulcerative colitis subjects to receive placebo orally single dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-3504 — TD-3504
  Arms: TD-3504 High-Dose; TD-3504 Low-Dose; TD-3504 Mid-Dose
Drug: 15N2-tofacitinib — 15N2-tofacitinib
  Arms: TD-3504 High-Dose; TD-3504 Low-Dose; TD-3504 Mid-Dose
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of single-dose TD-3504 and single dose 15N2-tofacitinib in healthy subjects and subjects with UC. The relative bioavailability of tofacitinib released from TD-3504 compared to co-administered oral heavy-labeled tofacitinib (15N2-tofacitinib) will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 to 55 years old
* Male subjects must abstain from sexual intercourse or use a highly effective method of birth control
* Women of child bearing potential must have a negative pregnancy test and either abstain from sex or use a highly effective method of birth control
* Body Mass Index (BMI) 18 to 32 kg/m2
* Willing and able to give informed consent
* Additional inclusion criteria apply

Inclusion Criteria for Ulcerative Colitis (UC) subjects:

* Subject has a history of UC
* Subject is either not taking any medication for UC or has been taking a stable dose of ulcerative colitis medications for ≥ 14 days
* Additional inclusion criteria apply

Exclusion Criteria:

* Is positive for hepatitis A, B or C, HIV or tuberculosis
* Has clinically significant abnormalities in baseline laboratory evaluations
* Subject has a clinically significant abnormal electrocardiogram (ECG)
* Participated in another clinical trial of an investigational drug (or medical device) within 30 days prior to screening (or within 60 days prior to screening if investigational drug was a biologic, or is currently participating in another trial of an investigational drug (or medical device)
* Additional exclusion criteria apply

Exclusion Criteria for Healthy Subjects:

* Use of prescription drugs or any chronic over the counter medications within 14 days prior to clinic admission or requires continuing use during study participation, with the exception of hormonal contraceptives or hormone replacement therapy or standard daily multivitamin.
* Additional exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability of TD-3504 by assessing the number, severity, and type of adverse events | Day 1 through Day 8
  To assess the safety & tolerability of TD-3504 following single escalating doses of TD-3504 co-administered with a low dose of 15N2 tofacitinib for 8 days in healthy subjects and subjects with UC by assessing the number, severity, and type of treatment related adverse events.

SECONDARY OUTCOMES:
Safety & tolerability of TD-3504 by assessing treatment related changes safety laboratory values | Day 1 through Day 8
  To assess the safety & tolerability of TD-3504 following single escalating doses of TD-3504 co-administered with a low dose of 15N2 tofacitinib for 8 days in healthy subjects and subjects with UC by assessing treatment related changes safety laboratory values.
Systemic area under the curve of TD-3504 | Day 1 through Day 4
  To assess the systemic exposure of TD-3504 following single escalating doses of TD-3504 and co-administered 15N2-tofacitinib.
Systemic Cmax of TD-3504 | Day 1
  To assess the systemic exposure of TD-3504 following single escalating doses of TD-3504 and co-administered 15N2-tofacitinib.
Systemic area under the curve of tofacitinib | Day 1 through Day 4
  To assess the systemic exposure of tofacitinib following single escalating doses of TD-3504 and co-administered 15N2-tofacitinib.
Systemic Cmax of tofacitinib | Day 1
  To assess the systemic exposure of tofacitinib following single escalating doses of TD-3504 and co-administered 15N2-tofacitinib.
Systemic area under the curve of 15N2-tofacitinib | Day 1 through Day 4
  To assess the systemic exposure of following single escalating doses of TD-3504 and co-administered 15N2-tofacitinib.
Systemic Cmax of 15N2-tofacitinib | Day 1
  To assess the systemic exposure of following single escalating doses of TD-3504 and co-administered 15N2-tofacitinib.
Tofacitinib relative bioavailability by area under the curve comparison | Day 1 through Day 4
  To assess the relative bioavailability of tofacitinib from TD-3504 relative to 15N2-tofacitinib.
Tofacitinib relative bioavailability by Cmax comparison | Day 1
  To assess the relative bioavailability of tofacitinib from TD-3504 relative to 15N2-tofacitinib.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.